CLINICAL TRIAL: NCT01108874
Title: Up-Down Determination of the ED90 of Metaraminol to Treat Hypotension During Elective Cesarean Section
Brief Title: Up-Down Determination of the ED90 of Metaraminol to Treat Hypotension During Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Jefferson Clivatti, MD, Disciplina de Anestesiologia, Universidade Federal de São Paulo
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: CEP1241/09
Record Dates: First submitted 2010-04-19; First posted 2010-04-22 (Estimated); Last update posted 2010-10-01 (Estimated); Status verified 2010-09

CONDITIONS: Hypotension
Keywords: Cesarean section; Hypotension; Metaraminol; Vasoconstrictor Agents; Adult; Female; Pregnancy; Anesthesia, Obstetrical/adverse effects; Anesthesia,Spinal; Blood Pressure/drug effects; Nausea; Vomiting
MeSH Terms: conditions — Hypotension; Nausea; Vomiting | interventions — Metaraminol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Metaraminol — Patients will be given metaraminol every time SBP falls below baseline value.

SUMMARY:
The purpose of this study is to find the best dose of metaraminol to be used in patients during elective cesarean sections.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effective dose 90% (ED90) of metaraminol to treat hypotension after spinal anesthesia in elective cesarean sections (CS). It is a double-blind study that uses the biased-coin up-down sequential allocation method to determine the ED90 of metaraminol.

Baseline systolic blood pressure (SBP) will be determined by three automated measures 3 minutes apart just before CS. During the period from induction of spinal anesthesia to fetal delivery SBP will be monitored every minute and metaraminol will be administered every time it is lower than baseline value. If SBP falls below 80% of baseline value, the treatment will be considered a failure. An adequate response will be defined as the absence of hypotension during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Elective CS under spinal anesthesia
* Normal singleton pregnancy beyond 36 weeks gestation
* ASA physical status I/II
* Age over 18 years

Exclusion Criteria:

* Patient refusal
* Allergy to metaraminol
* Preexisting or pregnancy-induced hypertension
* Cardiovascular or cerebrovascular disease
* Fetal abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The ED90 of Metaraminol to treat hypotension in elective cesarean section will be determined. | From spinal induction until delivery (on average 30-60min)
  Bolus doses of metaraminol will be used every time SBP falls below baseline values and maternal responses to doses will be used to build a dose response curve from where ED90 will be estimated.

SECONDARY OUTCOMES:
Maternal Demographics (Age, Height, Weight and Gestational Age)
Incidence of Nausea and Vomiting | From spinal induction until delivery (on average 30-60min)
Time between skin incision and delivery
Time between uterine incision and delivery
Total dose of metaraminol
Number of Participants with Hypertension or Bradycardia as a Measure of Safety and Tolerability | From spinal induction until delivery (on average 30-60min)
Umbilical blood gases
Fetal well-being with Apgar scores

CONTACTS AND LOCATIONS:
Overall Officials: Jefferson Clivatti, MD, Principal Investigator — Disciplina de Anestesiologia, UNIFESP
Locations (1):
- Hospital São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Tanaka M, Balki M, Parkes RK, Carvalho JC. ED95 of phenylephrine to prevent spinal-induced hypotension and/or nausea at elective cesarean delivery. Int J Obstet Anesth. 2009 Apr;18(2):125-30. doi: 10.1016/j.ijoa.2008.09.008. Epub 2009 Jan 21. PMID 19162468
- [Background] Pace NL, Stylianou MP. Advances in and limitations of up-and-down methodology: a precis of clinical use, study design, and dose estimation in anesthesia research. Anesthesiology. 2007 Jul;107(1):144-52. doi: 10.1097/01.anes.0000267514.42592.2a. PMID 17585226
- [Background] Ngan Kee WD, Lau TK, Khaw KS, Lee BB. Comparison of metaraminol and ephedrine infusions for maintaining arterial pressure during spinal anesthesia for elective cesarean section. Anesthesiology. 2001 Aug;95(2):307-13. doi: 10.1097/00000542-200108000-00009. PMID 11506099
- [Background] Ngan Kee WD, Lee A. Multivariate analysis of factors associated with umbilical arterial pH and standard base excess after Caesarean section under spinal anaesthesia. Anaesthesia. 2003 Feb;58(2):125-30. doi: 10.1046/j.1365-2044.2003.02888.x. PMID 12562407